CLINICAL TRIAL: NCT04305665
Title: HIV Study on MEasuring the Reservoir on Cellular Level to CUre Infection
Acronym: HIV-Mercuri
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-07056
Record Dates: First submitted 2020-02-21; First posted 2020-03-12 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Hiv
Keywords: HIV; Latency; Latency reversing agents; Latency reversal
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIV-1 positive persons

SUMMARY:
The aim of this study is to gain new insights into HIV latency and reversal through extensive blood and tissues sampling (lymph node and colon biopsies) from 25 individuals under ART.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 subtype B infection
* Able and willing to provide written informed consent
* Age = or >18 years and < 65 years
* CD4 count at screening > 350/μl
* Viral load < 40 copies/ml determined by CobasTaqMan HIV-1 test v2.0 assay for at least 2 years (one blip < 200 copies/ml is allowed)
* Ability and willingness to have blood and tissue samples collected and stored for 20 years and used for various research purposes.

Exclusion Criteria:

* Previous or current history of opportunistic infection (AIDS defining events as defined in category C of the CDC clinical classification), consisting of chronic HIV-1 infection.
* Evidence of active HBV infection (Hepatitis B surface antigen positive or HBV viral load positive in the past and no evidence of subsequent seroconversion (=HBV antigen or viral load negative and positive HBV surface antibody)).
* Evidence of active HCV infection: HCV antibody positive result within 60 days prior to study entry with positive HCV viral load or, if the HCV antibody result is negative, a positive HCV RNA result within 60 days prior to study entry.
* Current or known history of cardiomyopathy or significant ischemic or cerebrovascular disease.
* Current or known history of cancer.
* History of HIV-related thrombocytopenia.
* Pregnancy or breastfeeding.
* Any conditions, including preexisting psychiatric and psychological disorders, which will in the opinion of the investigator interfere with the trial conduct or safety of the participant.
* Previous participation in a trial evaluating an immune modulating agent.
* Abnormal results of standard of care laboratory tests:

  1. Confirmed haemoglobin <11g/dl for women and <12 g/dl for men
  2. Confirmed platelet count <100 000/µl *
  3. Confirmed neutrophil count <1000/μl
  4. Confirmed AST and/or ALT >10xULN
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Acute or serious illness, in the opinion of the site investigator, requiring systemic treatment and/or hospitalization within 60 days prior to entry.
* The following treatment will be prohibited three months before screening and during the study:

  1. immunosuppressive drugs (inclusive corticosteroids) except for drugs used for topical use.
  2. Immunomodulatory drugs including but not limited to Granulocyte-colony stimulating factors, Granulocyte-monocyte colony-stimulating factor, interleukin 2, 7 & 15.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-1 positive persons
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2020-06-24 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Quantification of HIV DNA and RNA | 5 years
  Digital PCR
Integration site analysis | 5 years
  HIV/host DNA junctions will be amplified using the Integration Site Loop Amplification (ISLA) assay, and resulting chimeric amplicons will be sequenced by Sanger.
Full-length HIV genome analysis | 5 years
  Full-Length Individual Proviral Sequencing (FLIPS) assay: nested PCR with Illumina MiSeq.
Epigenetic analysis | 5 years
  Methylation (bisulfite conversion) and chromatin accessibility (Assay for Transposase-Accessible Chromatin using sequencing)
Transcriptome analysis | 5 years
  * Bulk RNA sequencing on extracted RNA (Illumina Hiseq 2500 with 10-100 ng input of ribodepleted RNA)
  * Single cell RNA sequencing (10x genomics technology )
High dimensional phenotyping | 5 years
  CyTOF (mass cytometry, Fluidigm) combined with bioinformatics approach to extensively characterize the phenotype of latently infected cells
Immunohistochemistry, RNA- and DNA In Situ Hybridization | 5 years
  Immunochemistry will be used to study the expression of activation and exhaustion markers on tissues samples , while viral expression will be assessed through DNAScope and RNAScope technologies
Extracellular vesicles analysis | 5 years
  Extracellular vesicles (EV) will be isolated through size-exclusion chromatography (SEC) and Optiprep density gradient (ODG). The isolated EVs will be visualized by microscopy, western blot and PCR. Proteomics and RNA sequencing will be performed to assess the EV content.
Immunometabolic profile analysis | 5 years
  Mass spectrometry metabolomics will be used to study the immunometabolic profile of latently infected cells
p24 quantification | 5 years
  p24 SIMOA assay: ultra-sensitive digital immunoassay providing 1000 times improvement in detection limits compared with a traditional ELISA. This assay will be used to assess the capacity of various latency reversing agents and immunomodulators at reactivating HIV from latency.
Detection of translation-competent reservoirs | 5 years
  HIV-Flow assay: flow cytometry based assay using a combination of 2 antibodies targeting the p24 protein and allowing the detection of cells containing translation-competent viruses. p24+ cells detected by this assay can be sorted for downstream applications and further characterization of translation-competent reservoirs.

CONTACTS AND LOCATIONS:
Overall Officials: Linos Vandekerckhove, MD PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- [Derived] Delporte M, Lambrechts L, Blomme EE, van Snippenberg W, Rutsaert S, Verschoore M, De Smet E, Noppe Y, De Langhe N, De Scheerder MA, Gerlo S, Vandekerckhove L, Trypsteen W. Integrative Assessment of Total and Intact HIV-1 Reservoir by a 5-Region Multiplexed Rainbow DNA Digital PCR Assay. Clin Chem. 2025 Jan 3;71(1):203-214. doi: 10.1093/clinchem/hvae192. PMID 39749517